CLINICAL TRIAL: NCT02191072
Title: Efficacy and Safety of Omalizumab in Patients With Severe Acute Urticaria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201404056MIPC
Record Dates: First submitted 2014-07-09; First posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Urticaria
Keywords: urticaria,omalizumab
MeSH Terms: conditions — Urticaria | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- omalizumab (Experimental): omalizumab 300mg subcutaneously once
  Interventions: Drug: omalizumab

INTERVENTIONS:
Drug: omalizumab — a recombinant DNA-derived humanized IgG1k monoclonal antibody that specifically binds to free human immunoglobulin E (IgE)
  Other Names: xolair

SUMMARY:
Efficacy of omalizumab in chronic spontaneous urticaria had been demonstrated in phase II and phase III studies. Clinical symptoms and signs had been significantly reduced with omalizumab as doses of 150 mg and 300 mg at 4-week intervals in patients with chronic spontaneous urticaria who remained symptomatic despite antihistamine treatment. Omalizumab had an onset of effect within a week after initiation. Thus, the investigators hypothesize that omalizumab will be effective in the treatment of severe acute urticaria as add on therapy with a fast onset of action. Objective:To investigate the efficacy and safety of omalizumab in the treatment of severe acute urticaria Study design: This prospective, interventional, single-arm open label study will recruit patients with severe acute urticaria from emergency departments, hospitalized and outpatient departments. The included patients will receive a single subcutaneous dose of 300mg omalizumab therapy. The efficacy of omalizumab will be evaluated by physical examination and assessed by Urticaria Activity Score (UAS) at baseline, 1 hour, Day 1, Day3, Day 7, and 6 weeks after omalizumab therapy. The frequency and severity of treatment-emergent adverse events will also be evaluated

DETAILED DESCRIPTION:
Acute urticaria is defined as hives that persist less than 6 weeks. Some patients with acute urticaria may progressed and need urgent management at urgent care clinics and emergency rooms. Nonsedating H1-antihistamines represent the mainstay and corticosteroids and various immunosuppressive therapies are being used in severely affected patients, or for those patients who experience a poor response to antihistamines. However, even though already treated by antihistamines, the symptoms still last longer than 3 days in more than 34% of the patients. Efficacy of omalizumab in chronic spontaneous urticaria had been demonstrated in phase II and phase III studies. Clinical symptoms and signs had been significantly reduced with omalizumab as doses of 150 mg and 300 mg at 4-week intervals in patients with chronic spontaneous urticaria who remained symptomatic despite antihistamine treatment. Omalizumab had an onset of effect within a week after initiation. Thus, the investigators hypothesize that omalizumab will be effective in the treatment of severe acute urticaria as add on therapy with a fast onset of action. Objective:To investigate the efficacy and safety of omalizumab in the treatment of severe acute urticaria Study design: This prospective, interventional, single-arm open label study will recruit patients with severe acute urticaria from emergency departments, hospitalized and outpatient departments. The included patients will receive a single subcutaneous dose of 300mg omalizumab therapy. The efficacy of omalizumab will be evaluated by physical examination and assessed by Urticaria Activity Score (UAS) at baseline, 1 hour, Day 1, Day3, Day 7, and 6 weeks after omalizumab therapy. The frequency and severity of treatment-emergent adverse events will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-75 years(2)Documented diagnosis of acute urticaria within 3 years
* Documented diagnosis of acute urticaria within 3 years
* Daily UAS at the beginning of study more than or equal to 4
* At time of enrollment, the symptoms of this episode had persisted longer than 3 days even under oral/intravenous antihistamines with or without oral corticosteroid therapy

Exclusion Criteria:

* Weight < 20 kg
* Continuous use of suspected drugs that may induce acute urticaria
* Pregnant woman
* Evidence of parasitic infection defined as having the following three items:Risk factors for parasitic disease (living in an endemic area, chronic gastrointestinal (GI) symptoms, travel within the last 6 months to an endemic area and/or chronic immunosuppression) AND An absolute eosinophil count more than twice the upper limit of normal AND Evidence of parasitic colonization or infection on stool evaluation for ova and parasites. Note that stool ova and parasite evaluation will only be conducted in patients with both risk factors and an eosinophil count more than twice the upper limit of normal.
* Atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus or other skin disease associated with itch
* Treatment with omalizumab within 12 months before screening
* Treatment with any investigational agent within 30 days of screening
* IV immunoglobulin G (IVIG), or plasmapheresis within 30 days prior to Day -14
* Regular (daily/every other day) doxepin (oral) use within 6 weeks prior to Day -14
* Patients with current malignancy, history of malignancy, or currently under work-up for suspected malignancy except non-melanoma skin cancer that has been treated or excised and is considered resolved
* Hypersensitivity to omalizumab or any component of the formulation
* History of anaphylactic shock
* Presence of clinically significant cardiovascular, neurological, psychiatric, metabolic or other pathological conditions that could interfere with the interpretation of the study results and or compromise the safety of the patients
* Medical examination or laboratory findings that suggest the possibility of decompensation of co-existing conditions for the duration of the study. Any items that are cause for uncertainty must be reviewed with the Medical Monitor
* Inability to comply with study and follow-up procedures
* Evidence of current drug or alcohol abuse

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Change in daily Urticaria Activity Score | D0,1,2,3,4,5,6,7and 1 hour
  Change in daily UAS from baseline to Day7 in the treatment period

SECONDARY OUTCOMES:
Proportion of patient with daily UAS=0 at Day 1, Day 3 | Day 1,3
Change from baseline in itch severity score | Day 0,1,3
Change from baseline in size of largest hive score | Day 0,1, 3
Proportion of patient could stop H1-antihistamine treatment | Day 0,3
Proportion of angioedema-free days | Day 3,4,5,6,7
The frequency and severity of treatment-emergent AEs and SAEs | 6 weeks follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Tsai Tsen-Fang, Principal Investigator — Department of Dermatology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan